CLINICAL TRIAL: NCT01724281
Title: Outcome of Babies With Asymetry of Lateral Brain Ventricles
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0059-12
Record Dates: First submitted 2012-11-06; First posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Lateral Ventricles of Fetuses at Mid Trimester
Keywords: lateral ventricles; Asymetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — not relevant
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pregnant women between 19-30 weeks gestational age: No intervention, only follow up
  Interventions: Other: No intervention, only follow up

INTERVENTIONS:
Other: No intervention, only follow up

SUMMARY:
The investigators will follow up on babies that had prenatal diagnosis at 2nd or 3rd trimester of normal width and asymetry of lateral brain ventricles

DETAILED DESCRIPTION:
Women who will attend 2nd or 3rd ultrasound prenatal scans will be included. Women where the fetus would be diagnosed with lateral ventricles that are normal width (<10 m"m) but discrepacy of >3 m"m will be followed up after delivery by head ultrasound and neurologic exam

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women between 19-30 weeks gestational age and asymetry of lateral ventricles

Exclusion Criteria:

* Lateral ventricles >10 m"m

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women at 19-30 weeks who attend ultrasound exam and diagnosed with asymetry of lateral brain ventricles.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Lateral ventricles width after delivery | 2 years
  The investigators will follow up on brain ultrasound of babies with normal width discrepant lateral brain ventricles

SECONDARY OUTCOMES:
Neurologic examination of babies with discrepant but normal lateral ventricles | 2 years
  After delivery, a neurologic examination will be carried out on all babies with discrepant but normal lateral ventricles

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel